CLINICAL TRIAL: NCT05579080
Title: Predictive Factors for Failure of Non-invasive Ventilation and High-flow Oxygen Therapy in COVID-19 Patients: A Retrospective Observational Study.
Brief Title: Predictive Factors for Failure of Non-invasive Support Ventilation in Patients With COVID-19: A Retrospective Study.
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, JOSE ROBERTO LAPA E SILVA, Jose Roberto Lapa e Silva, Universidade Federal do Rio de Janeiro
Other Study IDs: 52534221.5.0000.5249
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pneumonia; COVID-19
Keywords: self-patient lung injury; outcome; COVID-19 infection; noninvasive ventilation
MeSH Terms: conditions — COVID-19 | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NIV group: group that performed only non-invasive ventilation
  Interventions: Device: noninvasive ventilation
- HFNC group: group that performed only oxygen therapy by high flow nasal cannula
  Interventions: Device: noninvasive ventilation
- NIV and HFNC group: group that used non-invasive ventilation and oxygen therapy by high flow nasal cannula
  Interventions: Device: noninvasive ventilation
- conventional oxygen therapy group: group that used only conventional oxygen therapy low-flow oxygen therapy.
  Interventions: Device: noninvasive ventilation

INTERVENTIONS:
Device: noninvasive ventilation — The medical records whose patients used some type of non-invasive ventilatory device and devices that promote oxygen supplementation will be analyzed.
  Other Names: conventional oxygen therapy; high flow nasal cannula

SUMMARY:
During the progression of COVID-19, some patients may require noninvasive ventilation (NIV) or high-flow nasal catheter (CNAF) oxygen therapy. The objective of the study is describe, retrospectively, possible predictor variables related to the use of NIV and CNAF, in order to associate them with their failure and consequent orotracheal intubation, through a retrospective analysis of a tertiary hospital in Rio de Janeiro. The primary and second outcomes are incidence of orotracheal intubation; time for OIT, length of stay in the ICU and hospital, and in-hospital mortality. The preliminary results shows that the absence of heart disease and dementia, as well as the acute onset of symptoms (less than or equal to 10 days) and age (between 40 and 79 years) showed a statistically significant trend.

DETAILED DESCRIPTION:
Introduction: COVID-19 is an infectious disease caused by SARS-CoV2 (severe acute respiratory syndrome by the novo coronavirus). During the progression of COVID-19 infection, some patients may require noninvasive ventilation (NIV) or high-flow nasal catheter oxygen therapy (HFNC). However, its use has proved controversial in this population. Objective: To describe, retrospectively, possible predictor variables related to the use of NIV and HFNC, in order to associate them with their failure and consequent orotracheal intubation. Materials and Methods: observational, retrospective study, according to STROBE model, from the analysis of medical records, between March 2020 and July 2021. Study approved by a co-substantiated committee of D'or research and teaching institute (CAAE: 52534221.5.0000.5249). Inclusion criteria: over 18 years of age, diagnosis of positive COVID-19, hospitalized in the ICU of a tertiary Hospital located in Rio de Janeiro, admitted between March 2020 and July 2021. Exclusion criteria: hospital stay time of less than 3 days; patients who evolved to IOT in less than 48 hours; patients whose therapy (NIV, CNAF or NIV + CNAF) lasted less than 48 hours; patients whose medical records do not have the variables for the study. Primary outcome: incidence of orotracheal intubation. Secondary outcomes: time for orotracheal intubation, length of stay in the ICU and hospital and in-hospital mortality. Statistical analysis: There was no sample calculation due to the exploratory, descriptive and retrospective nature of this study. The Mann-Whitney U test will be applied to assess differences in icu length of stay. Survival time as well as hospital length of stay until the event will be analyzed with Kaplan-Meier estimates; the log-rank test will be used for group comparison. The p-< 0.05 will be considered statistically significant. Preliminary results: 82.6% of the medical records completed phase 1 of data collection. Of these, 64.4% used CNAF, NIV or both. 20% of the medical records passed through phase 1 completed for phase 2 collection, with characterization of the population. The absence of heart disease and dementia, as well as the acute onset of symptoms (less than or equal to 10 days) and age (between 40 and 79 years) showed a statistically significant trend.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years of age and older,
* admitted to the ICU with COVID-19 confirmed by positive reverse transcriptase reaction followed by the polymerase chain reaction or chest CT suggestive of pneumonia caused by COVID-19
* admitted between March 2020 and July 2021.

Exclusion Criteria:

* Estimated length of hospital stay less than 3 days;

  * Patients who progressed to OTI in less than 48 hours of hospital stay;
  * Patients whose use of NIV and/or HFNC lasted less than 48 hours;
  * Patients whose medical records lack predictive and outcome variables.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients, 18 years of age and older, admitted to the ICU with COVID-19 confirmed by positive RT-PCR or chest CT suggestive of pneumonia caused by COVID-19, admitted between March 2020 and July 2021, who progressed to respiratory failure, requiring some ventilatory support or supplemental oxygen therapy
Sampling Method: Non-Probability Sample
Enrollment: 1319 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
orotracheal intubation | during hospitalization
  failure of noninvasive ventilatory therapy through the need for orotracheal intubation

SECONDARY OUTCOMES:
length of stay in the ICU | during hospitalization
  length of stay in the ICU
length of stay in hospital | during hospitalization
  length of stay in hospital
in-hospital mortality | during hospitalization
  in-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Silva, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (2):
- Brazil (2):
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - Barra D'or Hospital, Rio de Janeiro

REFERENCES:
- [Derived] da Cruz AP, Martins G, Martins CM, Marques V, Christovam S, Battaglini D, Robba C, Pelosi P, Rocco PRM, Cruz FF, Dos Santos Samary C, Silva PL. Comparison between high-flow nasal oxygen (HFNO) alternated with non-invasive ventilation (NIV) and HFNO and NIV alone in patients with COVID-19: a retrospective cohort study. Eur J Med Res. 2024 Apr 22;29(1):248. doi: 10.1186/s40001-024-01826-3. PMID 38649940

DOCUMENTS (1):
  • Study Protocol (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT05579080/Prot_000.pdf